CLINICAL TRIAL: NCT00239642
Title: Comparison of the Safety and Efficacy of Three Iron Sucrose Maintenance Regimens in Pediatric Chronic Kidney Disease (CKD) Patients
Brief Title: Safety and Efficacy of Iron Sucrose in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VEN03017
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2012-01-10 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Anemia; Chronic Kidney Disease
Keywords: Iron; Anemia; CKD
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Ferric Oxide, Saccharated

ARMS (3):
- Venofer (0.5 mg/kg) (Experimental): 0.5 mg/kg of Venofer (iron sucrose) up to 100 mg administered intravenously
  Interventions: Drug: Venofer (iron sucrose injection)
- Venofer (1.0 mg/kg) (Experimental): 1.0 mg/kg of Venofer (iron sucrose) up to 100 mg administered intravenously
  Interventions: Drug: Venofer (iron sucrose injection)
- Venofer (2.0 mg/kg) (Experimental): 2.0 mg/kg of Venofer (iron sucrose) up to 100 mg administered intravenously
  Interventions: Drug: Venofer (iron sucrose injection)

INTERVENTIONS:
Drug: Venofer (iron sucrose injection) — 0.5 mg/kg of Venofer (iron sucrose) up to 100 mg administered intravenously
  Arms: Venofer (0.5 mg/kg)
Drug: Venofer (iron sucrose injection) — 1.0 mg/kg of Venofer (iron sucrose) up to 100 mg administered intravenously
  Arms: Venofer (1.0 mg/kg)
Drug: Venofer (iron sucrose injection) — 2.0 mg/kg of Venofer (iron sucrose) up to 100 mg administered intravenously
  Arms: Venofer (2.0 mg/kg)

SUMMARY:
Comparison of three potential iron sucrose maintenance regimens in pediatric chronic kidney disease (CKD) patients

DETAILED DESCRIPTION:
Randomized, controlled, open label trial of pediatric CKD patients on stable erythropoietin (EPO) therapy. Patients will be followed for 12 weeks to assess safety (incidence of adverse events) and efficacy (clinical success)

ELIGIBILITY:
Inclusion Criteria:

* Patients between 2 to 21 years of age
* Patients on stable hemodialysis (HD) or peritoneal dialysis (PD) regimen for 3 months for ≥ 3 months
* Non-dialysis dependent (NDD) patients with glomerular filtration rate (GFR) <60
* Hemoglobin (Hgb) ≥ 11g/dL to ≤ 13.5g/dL
* Ferritin ≤ 800 ng/mL
* Transferrin saturation (TSAT) ≥ 20% to ≤ 50%
* Received stable erythropoietin (EPO) regimen for ≥ 8 weeks prior to the qualifying screening visit

Exclusion Criteria:

* Known hypersensitivity to iron sucrose
* Severe diseased of the liver, cardiovascular system, or hemopoietic system
* Serious infection requiring hospitalization
* Significant blood loss within the last 3 months
* Bleeding disorders
* Pregnancy / Lactation
* Actively being treated for asthma
* Hemoglobinopathy
* Receiving a myelosuppressive drug

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 141 (Actual)
Dates: Start 2005-07; Primary Completion 2009-01 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Falone, MD, Study Director — American Regent, Inc.
Locations (1):
- Luitpold Pharmaceutials, Norristown, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and Medical Clinics; Study Period - October 24, 2005 through January 23, 2009
Pre-assignment Details: Stable erythropoietin (EPO) dose (±25% of current dose) for 8 weeks prior to the qualifying screening visit.
Period: Overall Study
Arm/Group | Venofer (0.5 mg/kg) | Venofer (1.0 mg/kg) | Venofer (2.0 mg/kg)
Started | 49 | 47 | 49
Completed | 47 | 47 | 47
Not Completed | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Venofer (0.5 mg/kg) | Venofer (1.0 mg/kg) | Venofer (2.0 mg/kg) | Total
Number analyzed (Participants) | 49 | 47 | 49 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44 | 42 | 44 | 130
  Between 18 and 65 years | 5 | 5 | 5 | 15
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (4.40) | 13.1 (4.62) | 13.1 (4.87) | 13.3 (4.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 18 | 61
  Male | 28 | 25 | 31 | 84
Region of Enrollment [Number; unit: participants]
  United States | 26 | 31 | 25 | 82
  Russian Federation | 23 | 16 | 24 | 63

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile: Number of Subjects Experiencing at Least 1 Adverse Event
Description: Safety Profile: Number of subjects who experienced at least 1 adverse event in each arm
Time Frame: baseline through week 12
Population: Safety Population - Subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Venofer (0.5 mg/kg) | Venofer (1.0 mg/kg) | Venofer (2.0 mg/kg)
Number analyzed (Participants) | 47 | 47 | 47
participants | 27 | 25 | 26

2. Secondary Outcome: Number of Subjects Achieving Clinical Success
Description: Summary of the Number of Subjects Achieving Clinical Success During the 12-Week Study Period - Hemoglobin between 10.5 g/dL and 14.0 g/dL, Inclusive, TSAT between 20% and 50%, Inclusive, and Stable EPO Dosing (±25% of Baseline Dose)
Time Frame: anytime during the 12 week post-baseline period
Population: mITT subjects
Measure: Number; unit: participants
Arm/Group | Venofer (0.5 mg/kg) | Venofer (1.0 mg/kg) | Venofer (2.0 mg/kg)
Number analyzed (Participants) | 46 | 45 | 40
participants | 44 | 40 | 33

3. Secondary Outcome: Percentage (%) of Subjects Achieving Clinical Success
Description: Summary of the Percentage (%) of Subjects Achieving Clinical Success During the 12-Week Study Period - Hemoglobin between 10.5 g/dL and 14.0 g/dL, Inclusive, TSAT between 20% and 50%, Inclusive, and stable EPO Dosing (±25% of Baseline Dose)
Time Frame: anytime during the 12 week post-baseline period
Population: mITT subjects
Measure: Number; unit: percentage of subjects
Arm/Group | Venofer (0.5 mg/kg) | Venofer (1.0 mg/kg) | Venofer (2.0 mg/kg)
Number analyzed (Participants) | 46 | 45 | 40
percentage of subjects | 95.7 | 88.9 | 82.5

4. Secondary Outcome: Number of Subjects With Hemoglobin Between 10.5 g/dL and 14.0 g/dL, Inclusive
Description: Summary of the Number of Subjects with Hemoglobin between 10.5 g/dL and 14.0 g/dL, Inclusive
Time Frame: anytime during the 12-week post-baseline period
Population: mITT subjects
Measure: Number; unit: participants
Arm/Group | Venofer (0.5 mg/kg) | Venofer (1.0 mg/kg) | Venofer (2.0 mg/kg)
Number analyzed (Participants) | 46 | 45 | 40
participants | 46 | 43 | 38

5. Secondary Outcome: Percentage (%) of Subjects With Hemoglobin Between 10.5 g/dL and 14.0 g/dL, Inclusive
Description: Summary of the Percentage (%) of Subjects with Hemoglobin Between 10.5 g/dL and 14.0 g/dL, Inclusive
Time Frame: anytime during the 12 week post-baseline period
Population: mITT subjects
Measure: Number; unit: percentage of subjects
Arm/Group | Venofer (0.5 mg/kg) | Venofer (1.0 mg/kg) | Venofer (2.0 mg/kg)
Number analyzed (Participants) | 46 | 45 | 40
percentage of subjects | 100.0 | 95.6 | 95.0

6. Secondary Outcome: Proportion of Subjects With Transferrin Saturation (TSAT) Between 20% and 50%, Inclusive
Description: Summary of the Proportion of Subjects with transferrin saturation (TSAT) between 20% and 50%, Inclusive
Time Frame: anytime during the 12 week post-baseline period
Population: mITT subjects
Measure: Number; unit: participants
Arm/Group | Venofer (0.5 mg/kg) | Venofer (1.0 mg/kg) | Venofer (2.0 mg/kg)
Number analyzed (Participants) | 46 | 45 | 40
participants | 44 | 42 | 37

7. Secondary Outcome: Percentage (%) of Subjects With TSAT Between 20% and 50%, Inclusive
Description: Summary of the Percentage (%) of Subjects with TSAT between 20% and 50%, Inclusive
Time Frame: anytime during the 12 week post-baseline period
Population: mITT subjects
Measure: Number; unit: percentage of subjects
Arm/Group | Venofer (0.5 mg/kg) | Venofer (1.0 mg/kg) | Venofer (2.0 mg/kg)
Number analyzed (Participants) | 46 | 45 | 40
percentage of subjects | 95.7 | 93.3 | 92.5

8. Secondary Outcome: Proportion of Subjects With Stable Erythropoietin (EPO) Dosing or a Decrease >25% in EPO Dose From Baseline
Description: Summary of the Proportion of Subjects with Stable erythropoietin (EPO) Dosing or a Decrease >25% in EPO dose from Baseline
Time Frame: anytime during the 12 week post-baseline period
Population: mITT subjects
Measure: Number; unit: participants
Arm/Group | Venofer (0.5 mg/kg) | Venofer (1.0 mg/kg) | Venofer (2.0 mg/kg)
Number analyzed (Participants) | 46 | 45 | 40
participants | 46 | 45 | 39

9. Secondary Outcome: Percentage (%) of Subjects With Stable EPO Dosing or a Decrease >25% in EPO Dose From Baseline
Description: Summary of the Percentage (%) of Subjects with Stable EPO Dosing or a Decrease >25% in EPO Dose from Baseline
Time Frame: anytime during the 12 week post-baseline period
Population: mITT subjects
Measure: Number; unit: percentage of subjects
Arm/Group | Venofer (0.5 mg/kg) | Venofer (1.0 mg/kg) | Venofer (2.0 mg/kg)
Number analyzed (Participants) | 46 | 45 | 40
percentage of subjects | 100.0 | 100.0 | 97.5

ADVERSE EVENTS:
Time Frame: 3 years and 10 months
Arm/Group | Venofer (0.5 mg/kg) | Venofer (1.0 mg/kg) | Venofer (2.0 mg/kg)
Serious Adverse Events (participants affected / at risk) | 5/47 | 10/47 | 10/47
Other Adverse Events (participants affected / at risk) | 13/47 | 15/47 | 14/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venofer (0.5 mg/kg) (N=47) | Venofer (1.0 mg/kg) (N=47) | Venofer (2.0 mg/kg) (N=47)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (2)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (3)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Transplant (Surgical and medical procedures) | 3 (3) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Venofer (0.5 mg/kg) (N=47) | Venofer (1.0 mg/kg) (N=47) | Venofer (2.0 mg/kg) (N=47)
Blood pressure increased (Investigations) | 2 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Headache (Nervous system disorders) | 2 | 4 | 2
Peritonitis (Gastrointestinal disorders) | 0 | 3 | 2
Renal Transplant (Surgical and medical procedures) | 3 | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 4 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less